CLINICAL TRIAL: NCT06707597
Title: The Effects of Interaction Among Patients on Pain, Anxiety, and Comfort After Orthopedic Surgery
Brief Title: Patient Interaction Effects on Pain, Anxiety, and Comfort After Orthopedic Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Nursemin ÜNAL, Associate Professor, Ankara University
Other Study IDs: AEŞH-BADEK-2024-773
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Pain; Anxiety; Surgery
Keywords: pain; anxiety; comfort; orthopedic surgery; patient interaction
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Interaction Group: Patients who undergo the same surgical procedure on the same day and stay in the same room during the postoperative period will form this group.
  Interventions: Other: Patient Interaction Group
- Control group: Patients who undergo the same surgical procedure on the same day and stay in a single room during the postoperative period will form this group.

INTERVENTIONS:
Other: Patient Interaction Group — No interventions or procedures will be applied to the patients. To evaluate whether the pain, anxiety, and comfort of patients undergoing the same surgical procedure are influenced by each other, the average scale scores of patients in double and single rooms will be compared.
  Other Names: Control Group
  Groups: Patient Interaction Group

SUMMARY:
This study aims to evaluate the effects of interaction among patients on pain, anxiety, and comfort after orthopedic surgery.

DETAILED DESCRIPTION:
Surgical procedures can cause pain and anxiety in patients, affecting their comfort levels. Orthopedic surgeries, in particular, are associated with high pain levels. For example, common orthopedic procedures like total knee and hip replacement can cause patients to experience severe pain on the first-day post-surgery. In modern surgical practices, pain management requires the combined use of both pharmacological and non-pharmacological methods. Additionally, various stressors in the hospital environment-such as the sounds of medical devices and monitors, and crowded hospital rooms-can create extra stress for orthopedic patients, especially those with limited mobility. Another important factor is the interaction among patients in the same environment. The presence of another patient in the same room can affect not only environmental comfort but also, through "emotional contagion," the patient's emotional state. Emotional contagion is defined as the transfer of emotions from one person to another, and this interaction can trigger patients' pain and anxiety levels. Particularly, patients who have undergone similar surgical experiences may share each other's emotions empathetically, thereby increasing pain and anxiety. This study aims to examine the effects of patient interaction in the same room on pain, anxiety, and comfort in orthopedic patients.

The study population will consist of patients who undergo lower and upper extremity surgeries in the orthopedics and traumatology clinic of a state hospital in Turkey. Patients who undergo the same surgical procedure on the same day and stay in the same room postoperatively, or those who are in single rooms, will form the study sample. To obtain reliable results, at least 128 patients will be required, with 64 patients in the group sharing a room and 64 patients in the single-room control group. The goal is to reach this sample size during the planning and implementation phases of the research. Considering a 10% patient dropout rate, 70 patients in the shared room group and 70 patients in the single room group, for a total of 140 patients, will be included in the study. Patients will be grouped according to lower and upper extremity surgeries, and pairs will be formed for placement in the same rooms. Patients discharged within 24 hours will be evaluated during their hospital stay. Additionally, a control group of patients in single rooms will be included to assess the impact of staying in the same room.

Before surgery, the patients' trait anxiety levels will be measured using the State-Trait Anxiety Inventory. After the surgery, once patients are placed in their rooms, pain will be assessed at 1, 4, 8, 12, 16, and 24 hours using the Visual Analog Scale for pain at the surgical site, back, and head/neck. Also, at 1, 8, and 24 hours, their state anxiety and immobilization comfort will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To have undergone lower and upper extremity surgery at a state hospital,
* To be over 18 years of age,
* To stay in the hospital for at least one night,
* To agree to participate in the study.

Exclusion Criteria:

* Patients who undergo emergency surgical procedures,
* Patients with language barriers, learning difficulties, or cognitive diseases such as dementia that prevent them from completing the questionnaires,
* Patients with epidural or other catheters,
* Patients who do not wish to participate in the study will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of all adult patients who have undergone lower and upper extremity surgery at the relevant state hospital during the study period, meet the inclusion criteria, and voluntarily agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Change from Visual Analog Scale | Postoperative assessments will be carried out at 1, 4, 8, 12, 16, and 24 hours after surgery.
  Visual Analog Scale (VAS) is a standard scale used to assess the intensity of pain. Pain severity is represented by "No pain = 0" and "Worst pain = 10," and it is evaluated on a scale from 0 to 10.
Change from State Anxiety Scale | Postoperative assessments will be carried out at 1, 8, and 24 hours after surgery.
  Spielberger State-Trait Anxiety Inventory: The scale, developed by Spielberger in 1970, was validated in Turkish. The scale measures two dimensions of anxiety: State Anxiety and Trait Anxiety. The State Anxiety Scale consists of 20 items that describe how individuals feel at a specific moment under certain conditions, reflecting their emotions related to the situation they are in. The Trait Anxiety Scale consists of 20 items describing how individuals generally feel. In total, the scale includes 40 four-point Likert-type questions. The scale contains both direct and reverse-scored items. In the State Anxiety Scale, there are 10 reverse-scored items, and in the Trait Anxiety Scale, there are 7 reverse-scored items. The reverse-scored items in the State Anxiety Inventory are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The reverse-scored items in the Trait Anxiety Inventory are items 21, 26, 27, 30, 33, 36, and 39.
Change from Trait Anxiety Scale | Inpatient admission
  Spielberger State-Trait Anxiety Inventory: The scale, developed by Spielberger in 1970, was validated in Turkish. The scale measures two dimensions of anxiety: State Anxiety and Trait Anxiety. The State Anxiety Scale consists of 20 items that describe how individuals feel at a specific moment under certain conditions, reflecting their emotions related to the situation they are in. The Trait Anxiety Scale consists of 20 items describing how individuals generally feel. In total, the scale includes 40 four-point Likert-type questions. The scale contains both direct and reverse-scored items. In the State Anxiety Scale, there are 10 reverse-scored items, and in the Trait Anxiety Scale, there are 7 reverse-scored items. The reverse-scored items in the State Anxiety Inventory are items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20. The reverse-scored items in the Trait Anxiety Inventory are items 21, 26, 27, 30, 33, 36, and 39.
Change from Immobility Comfort Scale | Postoperative assessments will be carried out at 1, 8, and 24 hours after surgery.
  The scale developed by Hogan-Miller in 1995 was validated for Turkish in a group of patients immobilized due to lower extremity surgery. The Immobility Comfort Scale (ICS) is a 20-item scale using Likert-type response options. Each statement in the questionnaire has a Likert-type response ranging from 1 to 6, from "strongly disagree" to "strongly agree." The positive and negative items are mixed in the questionnaire. For positive items, the highest score (6 points) indicates the highest level of comfort, while the lowest score (1 point) indicates the lowest level of comfort. To calculate the total score of the questionnaire, the scores for the negative items are reverse-coded and added to the scores for the positive items. The minimum and maximum total scores in the questionnaire are 20 and 120 points, respectively. The average item score ranges from 1 to 6 and is determined by dividing the total score by the number of items in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nursemin Unal, Study Director — Ankara University

REFERENCES:
- [Background] Andersson V, Bergstrand J, Engstrom A, Gustafsson S. The Impact of Preoperative Patient Anxiety on Postoperative Anxiety and Quality of Recovery After Orthopaedic Surgery. J Perianesth Nurs. 2020 Jun;35(3):260-264. doi: 10.1016/j.jopan.2019.11.008. Epub 2020 Mar 5. PMID 32147278
- [Background] Spielberger, C. D. (2010). State-trait anxiety inventory. In The Corsini Encyclopedia of Psychology (pp. 1-1). Wiley.
- [Background] Öner, N, & LeCompte A. (1985). Durumluk-Sürekli Kaygı Envanteri El Kitabı. 2. Baskı. İstanbul: Boğaziçi üniversitesi Yayınları.
- [Result] Tosun B, Aslan O, Tunay S, Akyuz A, Ozkan H, Bek D, Aciksoz S. Turkish Version of Kolcaba's Immobilization Comfort Questionnaire: A Validity and Reliability Study. Asian Nurs Res (Korean Soc Nurs Sci). 2015 Dec;9(4):278-84. doi: 10.1016/j.anr.2015.07.003. Epub 2015 Sep 16. PMID 26724235
- [Result] Caliskan E, Aksoy N. The Relationship Between Preoperative Anxiety Level and Postoperative Pain Outcomes in Total Hip and Knee Replacement Surgery: A Cross-sectional Study. J Perianesth Nurs. 2025 Feb;40(1):76-82. doi: 10.1016/j.jopan.2024.03.010. Epub 2024 Jul 8. PMID 38980235
- [Result] Xu JJ, Tang XT, Fu WC, Zheng JX, Jiang LP, Zhou YW, Yang QN. "Adjacent Bed Effect" of Total Knee Arthroplasty Patients During the Perioperative Period. Pain Manag Nurs. 2024 Feb;25(1):88-92. doi: 10.1016/j.pmn.2023.09.003. Epub 2023 Oct 20. PMID 37867077